CLINICAL TRIAL: NCT05015829
Title: Diagnostic Impact of Low-dose Dobutamine Echocardiography in Low-flow Low-gradient Aortic Stenosis
Acronym: DALLAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Nils Sofus Borg Mogensen, Doctor, Odense University Hospital
Other Study IDs: S-20190058; 19/34844 (Other: Danish Data Protection Agency, Sourthern Denmark)
Record Dates: First submitted 2021-07-15; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Aortic Valve Stenosis; Valvular Stenosis; Valvular Heart Disease
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases | interventions — Echocardiography, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Classical low-flow low-gradient aortic stenosis: LVEF<50% SVi < 35.0 mL/m2 Aortic mean gradient < 40 mmHg AVA < 1.0 cm2.
  Interventions: Diagnostic Test: Dobutamine Stress Echocardiography
- Paradoxical low-flow low-gradient aortic stenosis: LVEF>50% SVi < 35.0 mL/m2 Aortic mean gradient < 40 mmHg AVA < 1.0 cm2.
  Interventions: Diagnostic Test: Dobutamine Stress Echocardiography

INTERVENTIONS:
Diagnostic Test: Dobutamine Stress Echocardiography — Change in echocardiographic 2D and doppler measurements during infusion with Dobutamine 5 µg/kg/min till max dosage of 20 µg/kg/min.

SUMMARY:
When aortic valve-area is <1.0cm2 and transvalvular mean-gradient is >40mmHg, the diagnosis of severe aortic stenosis (AS) is straightforward. However, some patients present with an apparently reduced valve-area, despite transvalvular-gradient <40mmHg; Low-flow, low-gradient aortic stenosis (LFLG AS). When a patient with LFLG AS also presents with LVEF <50%, guidelines recommends performing a Low-Dose Dobutamine-echocardiography (LDDE) to confirm true-severe AS. However, nearly 30% of patients with LFLG AS do not show an adequate respond to Dobutamine. More commonly, patients present with the combination of LFLG AS, despite LVEF≥50%. In this group of patients the use of LDDE remains undisclosed.

The purpose of this study is to examine the safety and diagnostic usefulness of LDDE in patients with LFLG AS with LVEF≥50%. Furthermore we will examine factors associated with inadequate response to LDDE.

150 symptomatic and/or asymptomatic patients with LFLG and LVEF≥50% and a control group with LVEF<50% will be enrolled at the Department of Cardiology, OUH. Patients will undergo clinical evaluation including LDDE, blood analyses, CT-scan and cardiac Mri.

Only a limited number of studies examine the possible use of LDDE in patients with LFLG AS and LVEF≥50% and no study has been performed documenting the safety and feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Low-flow (SVi<35 ml/m2) low-gradient (mean gradient <40 mmHg) AS with estimated AVA<1.0 cm2 referred to the Department of Cardiology, Odense University Hospital.
2. Age > 18 years.
3. Signed informed consent.

Exclusion Criteria:

1. Other moderate-severe valvular heart disease.
2. Unwilling to participate in the study.
3. Poor echocardiographic window.
4. Inability to follow-up due to temporary citizenship Registration Number (CPR-Number) or emigration within the study period.
5. Pregnant women.
6. Patients with severe chronic renal failure (eGFR<40 ml/min) will not undergo cardiac MRi or CT angiography.
7. Known contrast allergy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with LFLG AS followed at the Department of Cardiology, Odense University Hospital will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse effects during Dobutamine infusion | Dobutamine infusion, up to 30 minutes
  1. The occurrence of angina pectoris, severely high systolic blood pressure >200 mmHg or ventricular premature beats Lown Grade >3 or supra-ventricular arrhythmias or tachycardia assessed by ECG.
  2. Occurrence of signs of echocardiographic subvalvular obstruction; (systolic anterior motion of the mitral leaflet (SAM), high velocities (>2 m/sec) in the LV outflow tract and late peaking systolic jet).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  a) Gender (male/female).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  b) Aortic valve calcification assessed by cardiac CT (AU).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  c) Myocardial fibrosis assessed by MRi (%).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  d) Baseline myocardial systolic and diastolic function estimated by echocardiography (Global Longitudinal Strain (%), Strain Ratesystolic (SRs), deceleration time of mitral E-wave (ms) and end-systolic wall-stress corrected LVEF (dynes).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  e) The ongoing use of beta-blockers (%, dosis).
Factors associated with flow-reserve | Dobutamine infusion, up to 30 minutes
  f) Association with outcomes (rate of AVR, hospitalization for cardiac failure, death).
The ability of LDDE to predict outcome in patients with paradoxical low-flow, low-gradient aortic stenosis. | 1 day til 3 years
  Rate of AVR
The ability of LDDE to predict outcome in patients with paradoxical low-flow, low-gradient aortic stenosis. | 1 day til 3 years
  Hospitalization for cardiac failure
The ability of LDDE to predict outcome in patients with paradoxical low-flow, low-gradient aortic stenosis. | 1 day til 3 years
  All-cause mortality
The ability of LDDE to predict outcome in patients with paradoxical low-flow, low-gradient aortic stenosis. | 1 day til 3 years
  Cardiovascular mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Odense, Fune, Denmark

IPD SHARING:
Plan to Share IPD: Undecided